CLINICAL TRIAL: NCT05906225
Title: The Impact of Electroencephalogram (EEG) - Guided Inhalational Anesthetic Control on the Occurrence of EEG Discontinuity in Infants: A Prospective Randomized Controlled Trial
Brief Title: Anesthesia and EEG Discontinuity in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2304-138-1427
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia, General; Electroencephalography; Infant; Anesthesia, Inhalation
Keywords: Electroencephalography; Infant; General anesthesia; Burst suppression; Sevoflurane
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroencephalogram (Experimental): Adjustment of concentration of sevoflurane according to EEG
  Interventions: Procedure: EEG guided anesthesia
- Conventional (Active Comparator): Adjustment of concentration of sevoflurane according to vital signs
  Interventions: Procedure: Conventional anesthesia

INTERVENTIONS:
Procedure: EEG guided anesthesia — Monitoring of electroencephalogram via Sedline probe by MASIMO corporation. Adjust concentration of inhalational sevoflurane during anesthesia, according to component of slow&delta wave and alpha wave, so that slow/delta oscillation (with or without alpha oscillation) is maintained.
  Arms: Electroencephalogram
Procedure: Conventional anesthesia — Adjust concentration of inhalational sevoflurane during anesthesia, according to vital signs, so that mean blood pressure and heart rate are maintained between 80% and 120% of baseline values measured at ward before anesthesia.
  Arms: Conventional

SUMMARY:
This study is a randomized controlled trial to evaluate whether EEG-guided calibration of inhalation agents can reduce occurrence of EEG discontinuity in infants during general anesthesia.

DETAILED DESCRIPTION:
This is a study for comparison of incidence of EEG discontinuity during general anesthesia using sevoflurane. EEG guidance group will receive calibration of fraction of inhalational sevoflurane according to components of slow wave and delta wave of raw EEG. Control group will receive conventional management of anesthesia according to vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Infants who were born as full-term (>37 weeks postconception) and are equal to or less than 12 month old who were scheduled to undergo surgery under general anesthesia using inhalation agents.
* Belongs to American Society of Anesthesiologists Physical Status 1 or 2

Exclusion Criteria:

* Infants who were born less than 37 weeks postconception or has history of mechanical ventilation immediately after birth
* Presence of any genetic disease, chromosomal anomaly or congenital anomaly that can affect brain development
* Presence of any disease or disability in central nervous system
* History of trauma at head or surgery on brain
* History of hypersensitivity to any anesthetic agents
* Status of sedation or endotracheal intubation before induction of anesthesia
* Inability to attach probes for EEG monitoring
* Expectation of operation time as less than 5 minutes
* Other conditions that researchers regard as inappropriate for enrollment

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
EEG discontinuity | From start of anesthesia to end of anesthesia, Less than 24 hours
  Incidence of EEG discontinuity (EEG amplitudes < 25uV for more than 2 seconds)

SECONDARY OUTCOMES:
Total duration of EEG discontinuity | From start of anesthesia to end of study, Less than 24 hours
  Total sum of duration of EEG discontinuity
Significant isoelectric EEG | From start of anesthesia to end of study, Less than 24 hours
  Incidence of significant isoelectric EEG (EEG amplitudes < 10uV for more than 2 seconds)
EtSev | From start of anesthesia to end of study, Less than 24 hours
  Mean end-tidal sevoflurane concentration during anesthesia
SEF | From start of anesthesia to end of study, Less than 24 hours
  Mean spectral edge frequency value during anesthesia
PSi | From start of anesthesia to end of study, Less than 24 hours
  Mean patient state index value during anesthesia
Mean blood pressure | From start of anesthesia to end of study, Less than 24 hours
  Mean blood pressure values during anesthesia measured every 2.5 minutes
Heart rate | From start of anesthesia to end of study, Less than 24 hours
  Heart rate values during anesthesia measured every 2.5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hyun Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Other, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornelissen L, Kim SE, Purdon PL, Brown EN, Berde CB. Age-dependent electroencephalogram (EEG) patterns during sevoflurane general anesthesia in infants. Elife. 2015 Jun 23;4:e06513. doi: 10.7554/eLife.06513. PMID 26102526
- [Background] Cornelissen L, Kim SE, Lee JM, Brown EN, Purdon PL, Berde CB. Electroencephalographic markers of brain development during sevoflurane anaesthesia in children up to 3 years old. Br J Anaesth. 2018 Jun;120(6):1274-1286. doi: 10.1016/j.bja.2018.01.037. Epub 2018 Apr 5. PMID 29793594
- [Background] Tokuwaka J, Satsumae T, Mizutani T, Yamada K, Inomata S, Tanaka M. The relationship between age and minimum alveolar concentration of sevoflurane for maintaining bispectral index below 50 in children. Anaesthesia. 2015 Mar;70(3):318-22. doi: 10.1111/anae.12890. Epub 2014 Oct 1. PMID 25271891
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Bong CL, Long MHY. Sevoflurane requirements during electroencephalogram (EEG)-guided vs standard anesthesia care in children: A randomized controlled trial. J Clin Anesth. 2023 Jun;86:111071. doi: 10.1016/j.jclinane.2023.111071. Epub 2023 Feb 13. No abstract available. PMID 36774668
- [Background] Pawar N, Barreto Chang OL. Burst Suppression During General Anesthesia and Postoperative Outcomes: Mini Review. Front Syst Neurosci. 2022 Jan 7;15:767489. doi: 10.3389/fnsys.2021.767489. eCollection 2021. PMID 35069132
- [Background] Yuan I, Landis WP, Topjian AA, Abend NS, Lang SS, Huh JW, Kirschen MP, Mensinger JL, Zhang B, Kurth CD. Prevalence of Isoelectric Electroencephalography Events in Infants and Young Children Undergoing General Anesthesia. Anesth Analg. 2020 Feb;130(2):462-471. doi: 10.1213/ANE.0000000000004221. PMID 31107263
- [Background] Gao Z, Zhang J, Wang X, Yao M, Sun L, Ren Y, Qiu D. A retrospective study of electroencephalography burst suppression in children undergoing general anesthesia. Pediatr Investig. 2021 Aug 16;5(4):271-276. doi: 10.1002/ped4.12287. eCollection 2021 Dec. PMID 34938968
- [Background] Cornelissen L, Bergin AM, Lobo K, Donado C, Soul JS, Berde CB. Electroencephalographic discontinuity during sevoflurane anesthesia in infants and children. Paediatr Anaesth. 2017 Mar;27(3):251-262. doi: 10.1111/pan.13061. Epub 2017 Feb 8. PMID 28177176
- [Background] Yuan I, Xu T, Skowno J, Zhang B, Davidson A, von Ungern-Sternberg BS, Sommerfield D, Zhang J, Song X, Zhang M, Zhao P, Liu H, Jiang Y, Zuo Y, de Graaff JC, Vutskits L, Olbrecht VA, Szmuk P, Kurth CD; BRAIN Collaborative Investigators. Isoelectric Electroencephalography in Infants and Toddlers during Anesthesia for Surgery: An International Observational Study. Anesthesiology. 2022 Aug 1;137(2):187-200. doi: 10.1097/ALN.0000000000004262. PMID 35503999
- [Background] Katoh T, Kobayashi S, Suzuki A, Kato S, Iwamoto T, Bito H, Sato S. Fentanyl augments block of sympathetic responses to skin incision during sevoflurane anaesthesia in children. Br J Anaesth. 2000 Jan;84(1):63-6. doi: 10.1093/oxfordjournals.bja.a013384. PMID 10740549
- [Background] Avidan MS, Zhang L, Burnside BA, Finkel KJ, Searleman AC, Selvidge JA, Saager L, Turner MS, Rao S, Bottros M, Hantler C, Jacobsohn E, Evers AS. Anesthesia awareness and the bispectral index. N Engl J Med. 2008 Mar 13;358(11):1097-108. doi: 10.1056/NEJMoa0707361. PMID 18337600
- [Background] Lerman J, Sikich N, Kleinman S, Yentis S. The pharmacology of sevoflurane in infants and children. Anesthesiology. 1994 Apr;80(4):814-24. doi: 10.1097/00000542-199404000-00014. PMID 8024136
- [Background] Chao JY, Gutierrez R, Legatt AD, Yozawitz EG, Lo Y, Adams DC, Delphin ES, Shinnar S, Purdon PL. Decreased Electroencephalographic Alpha Power During Anesthesia Induction Is Associated With EEG Discontinuity in Human Infants. Anesth Analg. 2022 Dec 1;135(6):1207-1216. doi: 10.1213/ANE.0000000000005864. Epub 2022 Nov 16. PMID 35041633
- [Background] Lee HC, Jung CW. Vital Recorder-a free research tool for automatic recording of high-resolution time-synchronised physiological data from multiple anaesthesia devices. Sci Rep. 2018 Jan 24;8(1):1527. doi: 10.1038/s41598-018-20062-4. PMID 29367620